CLINICAL TRIAL: NCT04857840
Title: A Phase 3, Double-blind, Placebo-controlled and Open-label Efficacy and Long-term Safety Study of Firibastat (QGC001) Administered Orally, Once Daily, for Up to 48 Weeks in Patients With Difficult-to-treat/Resistant Hypertension.
Brief Title: Randomized Study of Extended Treatment With Firibastat in Treatment-Resistant Hypertension (REFRESH)
Acronym: REFRESH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No Efficacy demonstrated inn the QGC001-3QG1 study
Sponsor: Quantum Genomics SA (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QGC001-3QG2
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Hypertension (HTN)
MeSH Terms: conditions — Hypertension | interventions — firibastat

STUDY DESIGN:
Intervention Model Description: 2 Arms : Double-blind placebo controlled during Period 1 of 12 weeks followed by open-label periods 2 (24 weeks) and 3 (12 weeks)
Who Masked: Participant, Care Provider
Masking Description: Random allocation of the double blinded 2 Arms : Double-blind placebo controlled during Period 1 of 12 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Investigational Product /Period 1,2 and 3 if any (open label) (Experimental): Firibastat 1000 mg tablets QD - 12 weeks
  Interventions: Drug: Firibastat (QGC001) Period 1
- Arm B: Placebo/Period1 only (Placebo Comparator): Placebo tablets QD 12 weeks in Period 1 only, followed by open label Period 2 and 3 if any.
  Interventions: Drug: Firibastat (QGC001) Period 1

INTERVENTIONS:
Drug: Firibastat (QGC001) Period 1 — 1000 mg (2 x 500 mg) tablets QD per Os
  Other Names: Firibastat (QGC001) Open label

SUMMARY:
This is a double-blind, placebo-controlled and open-label, multicenter efficacy and long-term safety study of firibastat (QGC001) 1000 mg (2×500 mg tablets) administered po, QD, for up to 48 weeks in patients with difficult-to-treat/treatment-resistant HTN. Subjects will continue to take their chronic antihypertensive therapies (at least 2 classes of antihypertensive therapies) at the MTDs during the Run in Period and for the duration of the study. For treatment-resistant subjects, one of the antihypertensive therapies must be a diuretic; for difficult-to-treat subjects, the antihypertensive therapies do not have to include a diuretic. Subjects will complete subject medication diaries during the Run-in Period. If systolic automated office BP (AOBP) is ≥180 mmHg or diastolic BP (DBP) ≥110 mmHg at any visit during the study (and repeated and confirmed within 30 min), the subject will be withdrawn from the study and will receive appropriate treatment.

DETAILED DESCRIPTION:
For each subject, the study will include a Screening Visit, a Run-in Period, an Inclusion Visit (Visit 2A, Day 0, and Visit 2B, Day 1), and up to 3 study treatment periods with clinic visits and safety phone calls.

Screening assessments will be performed at Visit 1, Day -28. Eligible subjects will then enter the Run-in Period, during which medication adherence will be assessed via a medication diary. The duration of the Run in Period will be no less than 28 days and no more than 33 days; this time period allows for 2 repeat ambulatory BP monitoring (ABPM) recordings at Visit 2A, if required.

Subjects who meet the inclusion/exclusion criteria at the end of the Run in Period will be randomly assigned to either Group A or Group B. A total of 200 subjects (100 in Group A and 100 in Group B) will be randomized to continue treatment with firibastat (QGC001) during Period 3. Subjects will receive either double-blind firibastat (QGC001) or placebo for the first 12-week study treatment period (Period 1), followed by open label treatment with firibastat for 24 weeks (Period 2), or 36-weeks (Period 2 plus an additional 12-weeks of open-label treatment in Period 3).

At Visit 2A, Day 0, an ABPM device will be installed for each subject who has successfully completed the Run-in Period with a medication adherence ≥80%, and remains eligible to participate in the study. The ABPM device will be set to record for at least 24 hours, with the measurement frequency set at 30-minute intervals during the day (8:00 am to 10:00 pm [theoretically 28 readings, 2 per hour]) and 60-minute intervals at night (10:00 pm to 8:00 am [theoretically 10 readings, 1 per hour]). Subjects must have a successful ABPM measurement prior to being randomized and starting treatment with investigational product (IP) at Visit 2B, Day 1. An ABPM recording is considered successful if at least 21 daytime readings and 6 nighttime readings have been successfully recorded. A duration of less than 24 hours (e.g., 23 hours and 30 minutes) would be acceptable for a successful ABPM recording providing it successfully confirms 21 daytime readings and 6 nighttime readings. If the ABPM recording is not successful, 2 further attempts are permitted.

Following a successful ABPM recording (assessed at Visit 2B, Day 1), subjects who still meet the inclusion/exclusion criteria and who have a mean daytime systolic ambulatory blood pressure (ABP) >135 mmHg, will undergo visit-specific assessments and will be randomized to Group A or Group B, and receive either firibastat (QGC001) or placebo for the 12-week double-blind treatment period (Period 1), followed by open label firibastat for 24 weeks (Period 2), or 36 weeks (Period 2 plus Period 3 [200 subjects]), in addition to their current chronic antihypertensive treatments.

During Period 1, the investigator (or designee) will call subjects by telephone on Day 14 (±3 d) to collect any potential adverse events (AEs), check IP compliance, and record any concomitant medications. Subjects will receive a second safety phone call during Period 2, at Day 98 (±3 d).

Subjects will attend the study site for the following study visits:

Period 1: Visit 2A, Day 0; Visit 2B, Day 1; Visit 3, Day 42 (±3 d); Visit 4A, Day 84 (±3 d); and Visit 4B, Day 85 (±3 d).

Period 2: Visit 5, Day 126 (±3 d); Visit 6, Day 168 (±3 d); Visit 7, Day 252 (±3 d); and Visit 8, Day 280 (±3 d).

Period 3:Visit 9, Day 336 (±3 d), and Visit 10, Day 364 (±3 d). On completion of their final study treatment period, subjects will attend an End of Treatment (EOT) Visit. A safety follow-up will be performed at the End of Study (EOS) Visit.

For subjects who stop study treatment at the end of Period 2, the EOT Visit will be at Visit 7, Day 252 (±3 d), and the EOS Visit will be Visit 8, Day 280 (±3 d).

Subjects who continue study treatment into Period 3 will not attend Visit 8, Day 280 (±3 d). Subjects who stop treatment with firibastat (QGC001) after Period 3 will attend an EOT Visit at Visit 9, Day 336 (±3 d), and an EOS Visit at Visit 10, Day 364 (±3 d).

Subjects who discontinue the study early should undergo an Early Termination Visit, and an EOS visit 28 days (±3 d) after the last dose of IP (except in the case of consent withdrawal).

Each subject will be assigned to one of 5 pharmacokinetic (PK) subgroups; 50 subjects (at selected sites) will undergo an enhanced PK sampling schedule (6 PK samples will be collected according to the PK subgroup sampling schedule), and 700 subjects will be assigned to the standard PK sampling schedule (2 PK samples will be collected according to the PK subgroup sampling schedule).

At each study visit, AOBP, orthostatic BP, and heart rate (HR) will be measured, and other visit-specific procedures will be performed, including electrocardiograms (ECGs), clinical laboratory evaluations, clinical examinations, collection of blood for PK samples and the biomarker N terminal pro-B-type natriuretic peptide (NT-ProBNP), and monitoring of AEs and concomitant medications. At the EOS Visit (safety follow-up) assessments will include clinical examination, AOBP, orthostatic BP, ECG, HR, and clinical laboratory assessments, AE monitoring, and concomitant medications.

Allergic skin reactions and/or diabetes insipidus (DI) are considered adverse events of special interest (AESIs) with immediate notification during the study treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to provide written informed consent, and able to comply with the study procedures and restrictions.
* Adult men and women (at Screening).
* Diagnosis of primary HTN for at least 6 months prior to Screening and:

  * Currently treated with 2 antihypertensive classes of drug (difficult-to-treat subjects), or currently treated with at least 3 antihypertensive classes of drug including a diuretic (treatment resistant subjects), at the MTDs of those medications (ie, the subject can tolerate the current dose of each medication but higher doses have caused or may worsen side effects), with no change in their antihypertensive regimen (drug, dose, or schedule) for at least 6 weeks, and with medication adherence ≥80% during the Run in Period.
  * Have a systolic AOBP between 140 mmHg and 179 mmHg (inclusive) at Screening while on their current chronic antihypertensive treatments.
  * Have a successful ABPM measurement with a mean systolic daytime ABP >135 mmHg after the Run-in Period while on their current chronic antihypertensive treatments. An ABPM is successful if at least 21 daytime readings and 6 nighttime readings have been successfully recorded.
* Women of childbearing potential and nonsurgically sterile male subjects who are sexually active must agree to use an approved highly effective form of contraception from the time of informed consent until 30 days post dose. Approved forms of contraception include hormonal intrauterine devices, hormonal contraceptives (oral birth control pills, depo, patch, or injectable) together with supplementary barrier methods such as condoms or diaphragms with spermicidal gel or foam.
* Women of childbearing potential must have a negative serum pregnancy test result at Screening and a negative urine pregnancy test result at the Inclusion Visit (Visit 2B, Day 1)

Exclusion Criteria:

* Target population:

Subjects with uncontrolled primary HTN despite being treated with at least 2 classes of antihypertensive therapies, at the MTDs (difficult-to-treat or treatment-resistant patients).

Inclusion criteria:

Subjects who meet all of the following criteria will be eligible to participate in the study:

1. Able to understand and willing to provide written informed consent, and able to comply with the study procedures and restrictions.
2. Adult men and women (at Screening).
3. Diagnosis of primary HTN for at least 6 months prior to Screening and:

   * Currently treated with 2 antihypertensive classes of drug (difficult-to-treat subjects), or currently treated with at least 3 antihypertensive classes of drug including a diuretic (treatment resistant subjects), at the MTDs of those medications (ie, the subject can tolerate the current dose of each medication but higher doses have caused or may worsen side effects), with no change in their antihypertensive regimen (drug, dose, or schedule) for at least 6 weeks, and with medication adherence ≥80% during the Run in Period.
   * Have a systolic AOBP between 140 mmHg and 179 mmHg (inclusive) at Screening while on their current chronic antihypertensive treatments.
   * Have a successful ABPM measurement with a mean systolic daytime ABP >135 mmHg after the Run-in Period while on their current chronic antihypertensive treatments. An ABPM is successful if at least 21 daytime readings and 6 nighttime readings have been successfully recorded.
4. Women of childbearing potential and nonsurgically sterile male subjects who are sexually active must agree to use an approved highly effective form of contraception from the time of informed consent until 30 days post dose. Approved forms of contraception include hormonal intrauterine devices, hormonal contraceptives (oral birth control pills, depo, patch, or injectable) together with supplementary barrier methods such as condoms or diaphragms with spermicidal gel or foam.
5. Women of childbearing potential must have a negative serum pregnancy test result at Screening and a negative urine pregnancy test result at the Inclusion Visit (Visit 2B, Day 1).

Exclusion criteria:

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Known or suspected secondary HTN (eg, hyperaldosteronism, renovascular HTN, pheochromocytoma, Cushing's disease).
2. Systolic AOBP ≥180 mmHg or DBP ≥110 mmHg at the Screening or Inclusion Visit (Visit 2B, Day 1) and confirmed by a second measurement within 30 minutes to 1 hour.
3. Known hypertensive retinopathy (Keith-Wagener Grade 3 or Grade 4) and/or hypertensive encephalopathy.
4. Upper arm circumference that is outside the limits of the study-provided BP cuff associated with either the ABPM and/or AOBP measurement device.
5. History of spontaneous or drug-induced angioedema.
6. History of any drug-related allergy or hypersensitivity to any components of the IP (firibastat [QGC001] or placebo).
7. Known severe aortic stenosis (symptomatic or asymptomatic with valvular indexed surface <0.5 cm²/m²).
8. Subjects with severe symptomatic heart failure (New York Heart Association [NYHA] Class III or Class IV).
9. History of acute coronary syndrome (non-ST elevation myocardial infarction [MI], ST elevation MI, and unstable angina pectoris), stroke, or transient ischemic attack within 6 months prior to Visit 2A, Day 0.
10. Known history of malabsorption syndrome, or has undergone gastrointestinal surgery, including bariatric procedures that induce chronic malabsorption, within 2 years of Screening.
11. Treatment with anti-obesity drugs or procedures 3 months prior to Screening (ie, surgery, aggressive diet regimen, etc.), leading to unstable body weight.
12. Female who is breastfeeding, pregnant, or planning to become pregnant during the study period.
13. Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 3 years.
14. Shift workers who routinely sleep during the daytime and/or whose work hours include midnight.
15. Subjects with moderate to severe hepatic impairment (Child-Pugh A, B, or C); alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >3×upper limit of normal (ULN), or a total bilirubin ≥1.5×ULN (unless secondary to Gilbert's syndrome), or direct bilirubin >ULN in subjects with Gilbert's syndrome at Screening.
16. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2, as calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula (Levey AS, et al. 2009) at Screening.
17. History of any blood disorder, other than sickle cell trait, causing hemolysis or unstable red blood cells (eg, malaria, babesiosis, hemolytic anemia, thalassemia, sickle cell anemia).
18. Subjects with documented DI.
19. Subjects with Type 1 diabetes mellitus.
20. Subjects with Type 2 diabetes mellitus who:

    * Are poorly controlled, defined as glycosylated hemoglobin A1c (HbA1c) >9% at Screening; OR
    * Are taking short-acting insulin. Use of a stable dose [≥12 weeks prior to Screening] of the following medications, (or any combination of the following medications) is permitted: glucagon like peptide 1 analog, metformin, sulfonylurea, dipeptidyl peptidase-4 inhibitor, and single basal insulin, sodium glucose co-transporter 2 (SGLT2) inhibitors and pioglitazone.
21. Routine or anticipated treatment with any systemic corticosteroid. Use of topical, inhaled, intra articular or nasal corticosteroids is permitted.
22. Clinical evidence of thyroid disease, thyroid hormone therapy that is not stable ≥4 weeks prior to Screening, or a thyroid-stimulating hormone (TSH) level <0.75×lower limit of normal or >1.5×ULN at Screening.
23. History of alcohol or drug abuse (including opioid overuse/misuse) within the 3 months prior to Screening that would interfere with study participation or lead to decreased compliance to study procedures or IP intake in the investigator's opinion.
24. Participation in another clinical study involving an investigational drug within 30 days prior to Screening or plans to participate in another clinical study within 30 days of discontinuation of IP.
25. Any other condition that precludes adequate understanding, cooperation, and compliance with study procedures or any condition that could pose a risk to the subject's safety, as per the investigator's judgment.
26. Subjects with a life expectancy of less than 1 year per investigator's discretion.
27. Legal incapacity or limited legal capacity.
28. Previous participation in any clinical study with firibastat (QGC001).
29. Subjects with any history of documented allergic reactions or allergic diseases, with the exception of documented seasonal allergies (per the investigator's decision).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change from baseline in systolic AOBP at Week 12. | 12 weeks
  The main criterion will be analyzed with a mixed model with repeated measures (MMRM) at Week 6 (Day 42) and Week 12 (Day 84), with an unstructured matrix of covariance.

CONTACTS AND LOCATIONS:
Overall Officials: Georges GB BAKRIS, MD, Study Chair — AHA Comprehensive Hypertension Center University of Chicago Medical Center
Locations (2):
- Manassas Clinical Research Center, Manassas, Virginia, United States
- Canadian Phase Onward, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No